CLINICAL TRIAL: NCT04148495
Title: Intravenous Acetaminophen and Morphine Versus Intravenous Morphine Alone for Acute Pain in the Emergency Department: a Multicenter Randomized Controlled Double-blind Non-inferiority Trial
Brief Title: Intravenous Acetaminophen and Morphine Versus Intravenous Morphine Alone for Acute Pain in the Emergency Department
Acronym: ADAMOPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC19_0116
Record Dates: First submitted 2019-10-28; First posted 2019-11-01 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Pain Management
Keywords: Morphine; acetaminophen; Acute pain; Analgesics
MeSH Terms: conditions — Agnosia; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Morphine IV and the placebo of acetaminophen IV.
  Interventions: Drug: placebo of acetaminophen IV
- Control group (Active Comparator): Morphine IV and acetaminophen IV
  Interventions: Drug: acetaminophen IV

INTERVENTIONS:
Drug: placebo of acetaminophen IV — Mophine IV: Initial loading dose of 0.1 mg/kg (ensuring that the maximum dose of 10 mg is not exceeded) followed by bolus of 0.05 mg/kg every 10 minutes (taking care not to exceed the maximum dose of 5 mg) as reported by the recommandation of experts of the french society of urgency care.
  Placebo of acetaminophen IV: Sodium chloride 0.9%
  Arms: Treatment group
Drug: acetaminophen IV — Mophine IV: Initial loading dose of 0.1 mg/kg (ensuring that the maximum dose of 10 mg is not exceeded) followed by bolus of 0.05 mg/kg every 10 minutes ((taking care not to exceed the maximum dose of 5 mg) as reported by the recommandation of experts of the french society of urgency care.
  Acetaminophen IV: 1 g
  Arms: Control group

SUMMARY:
In emergency medicine, acute pain is a common reason for consultation. It is recommended that patients in moderate to severe pain should receive a combination of intravenous acetaminophen and morphine. However, the data are sparse to support this strategy. Thus, the purpose of our research is to test non-inferiority of IV morphine alone versus IV acetaminophen and morphine in a multicenter, randomized, controlled double blind trial in ED patients with moderate to severe acute pain.

DETAILED DESCRIPTION:
This study is designed to assess whether IV morphine alone is non inferior to combination IV acetaminophen and morphine for the management of moderate to severe pain in the ED. Numeric rating scale pain score will be compared between those who receive morphine alone and who will receive acetaminophen and morphine at 15, 30, 45 and 60 min post first injection.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* Moderate to severe acute pain, defined as a numeric rating scale score greater than or equal to 5.
* Conscious patient
* Clinical stability at the physician's discretion
* Patient able to talk and give a verbal assessment of his/her pain with the numerical verbal scale
* Out of guardianship and/or tutorship
* Affiliated to the social security plan.

Exclusion Criteria:

* Pregnancy and Breast-feeding
* Patient Unable to give numeric rating scale scores
* Patient with a weight strictly less than 50kg.
* acute pulmonary edema, acute respiratory failure
* Acute coronary syndrome or unbalanced ischemic heart disease in progress.
* Acute alcoholic intoxication.
* Patient who received morphine, or acetaminophen, or analgesic, or anti-inflammatory, for the current acute pain episode, within 8 hours prior to arrival at the emergencies
* No possibility of having venous access
* History of chronic pain during treatment.
* Allergy, intolerance or know contraindication to paracetamol or morphine or to an excipient.
* Renal or hepatic insufficiency.
* Association with buprenorphine, nalbuphine and pentazocine.
* Patient unable or unable to give written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Comparison of numeric rating scale pain scores between those who received morphine alone and who received combination of acetaminophen and morphine at 30 minutes. | 30 minutes
  The Numerical Pain Rating Scale measures the perception of pain intensity with an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Comparison of numeric rating scale pain scores between those who received morphine alone and who received the combination of acetaminophen and morphine at 10min, 20 min, 45 min and 60min. | 60 minutes
  The Numerical Pain Rating Scale measures the perception of pain intensity with an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Estimated cumulative dose of morphine in both arms at a dose -by-weight (mg/kg) dose during the first 30 minutes | 30 minutes
Frequency and intensity of adverse reactions: nausea, vomiting, respiratory failure, hypotension | through study completion, an average of 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Céline LONGO, Doctor, Principal Investigator — Nantes University Hospital
Locations (11):
- France (11):
  - Angers University Hospital, Angers
  - Bordeaux University Hospital, Bordeaux
  - Châteaubriant Hôspital, Châteaubriant
  - Grenoble University Hospital, Grenoble
  - La Roche-sur-Yon Hospital, La Roche-sur-Yon
  - Nancy University Hospital, Nancy
  - Nantes University Hospital, Nantes
  - Lariboisière University Hospital - APHP, Paris
  - La Pitié-Salpêtrière University Hospital, Paris
  - ROUEN University hospital, Rouen
  - CH Saint Nazaire, Saint-Nazaire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cattin G, Jenvrin J, Hardouin JB, Longo C, Montassier E. Intravenous acetaminophen with morphine versus intravenous morphine alone for acute pain in the emergency room: protocol for a multicenter, randomized, placebo-controlled, double-blinded study (ADAMOPA). Trials. 2022 Dec 15;23(1):1016. doi: 10.1186/s13063-022-06943-0. PMID 36522767